CLINICAL TRIAL: NCT03085823
Title: The All-comers Sirolimus-coated Balloon European Registry
Acronym: EASTBOURNE
Status: Completed | Type: Observational
Sponsor: Fatebenefratelli and Ophthalmic Hospital (Other)
Responsible Party: Principal Investigator, Bernardo Cortese, MD FESC, Fatebenefratelli and Ophthalmic Hospital
Other Study IDs: fbf001
Record Dates: First submitted 2016-11-29; First posted 2017-03-21 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Percutaneous Coronary Intervention; Angioplasty, Balloon, Coronary; Coronary Angioplasty, Transluminal Balloon; Arteriosclerosis, Coronary
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Sirolimus Coated Balloon

SUMMARY:
The purpose of this study is to observe and evaluate the performance of a Sirolimus-eluting Drug Coated Balloon for the treatment of any type of coronary lesions, including native vessel disease and in stent restenosis.

DETAILED DESCRIPTION:
The drug coated balloons (DCB) are one of the most promising innovations in the interventional cardiology field, and in some cases represent a valid alternative to stents. The numerous devices currently on the market, and the clinical results sometimes encouraging, sometimes less, have clearly shown that there is no "class" effect. The DCB so far available were conformed to elute only paclitaxel, an high lipophilicity drug with a narrow therapeutic window, cytotoxic at medium-high dosage.

The DCB allow the drug release without needing to implant prostheses in the coronary vessel; such prostheses (stents have been shown to be associated with an increased risk of thrombotic events, even years after implantation, caused by a non- healing of the vessel by the action of the drug itself or of the polymer, together with the presence of the metal of the stent . After a DCP angioplasty the absence of such implants, instead, ensures a quick recovery of the vessel function. Moreover, the absence of the prosthesis is particularly favorable in the case of small/medium diameter vessels, tortuous or severe calcific vessel, or for the treatment of in-stent restenosis.

In the Bello study, the DCB IN.PACT Falcon, has reached the non-inferiority expected (and also the superiority, not expected), against the same DES regarding the primary endpoint of late lumen loss (LLL) at the angiographic control. The results of this study, encouraging for the drug-eluting balloon technology, however, are tainted by a now obsolete technology, the use of an endpoint that supports the balloon (LLL), and the comparison with a DES that is no longer in trade and is objectively inferior to those used in 2016.

Several new generation DCB have been developed in the last years, with the aim of improving the paclitaxel release in the coronary wall, thus reducing the risk of restenosis. In addition, several improvements have involved the trackability and deliverability of these devices even in tortuous and small vessels . The latest generation DCB have several advantages compared to the old generation DCB: paclitaxel is layered with an inert support (matrix or carrier) using a multi-layer technology, improving both its release and the persistence in the vessel wall; furthermore, significant improvements have been made to address the poor deliverability of first generation balloons.

In 2016 the Magic Touch, a new type of DCB has obtained, first, the CE mark for marketing in Europe; it is characterized by eluting sirolimus, a drug with potent inhibitory effect on cell growth, but with low lipophilicity. For this reason, its ability to penetrate the wall of the vessel is limited, and so far it has not been possible to develop a device that would allow an effective release, despite the drug is now known for years in cardiology.

The purpose of this study is to evaluate the DCB Magic Touch performance in terms of efficacy and safety when used during coronary angioplasty, in a wide spectrum of coronary heart disease.

The primary objective of the study is to verify the rate of target vessel revascularization (TLR) at 12 months after implantation, both with new coronary angioplasty or coronary artery bypass graft.

Secondary objectives will be:

* angiographic success, defined as residual stenosis < 50% and TIMI 3 coronary flow; - procedural success, defined as angiographic success and absence of adverse cardiovascular events during initial hospitalization;
* major adverse cardiac events (MACE ), a composite endpoint of cardiac death, acute myocardial infarction and need for TLR at 6, 12, 24 and 36 months of implantation;
* every single element determining the MACE endpoint. This is a multicenter, prospective, spontaneous, observational, single-arm, clinical study, where will be enrolled patients with coronary artery disease and clinical indication for coronary angioplasty.

The indication for coronary angioplasty will be stable angina pectoris, silent ischemia or acute coronary syndrome (unstable angina or acute myocardial infarction).

Before participating all subjects will be informed about the study, including the possible risks and benefit, and will be asked to provide a written informed consent. Subjects will be instructed that may not meet the general criteria for inclusion or those angiographic, or that could satisfy at least one criterion for exclusion and therefore be excluded from the study (screening failure), even after informed consent.

ELIGIBILITY:
Inclusion Criteria:

* age at least 18
* patients with symptomatic coronary artery disease (including chronic stable angina, silent ischemia, acute coronary syndromes) with clinical indication to percutaneous coronary intervention.

Exclusion Criteria:

* patients with one or more of the following criteria: known (and untreatable) hypersensitivity or contraindication to Aspirin, Heparin, Clopidogrel, Prasugrel, Ticagrelor, Sirolimus, or a sensitivity to contrast media which cannot be adequately pre-medicated.
* patients enrolled in another trial.

Target lesion/vessel with any of the following characteristics:

* successful pre-dilatation not performed in the target lesion, or not efficacious (residual stenosis >50%);
* severe calcification of the target vessel, also proximal to the lesion;
* highly tortuous lesions which can impair access of device to treatment site.
* visible thrombus at lesion which is not treatable with aspiration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a clinical indication for PCI.
Sampling Method: Non-Probability Sample
Enrollment: 2123 (Actual)
Dates: Start 2016-09; Primary Completion 2020-12 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Target lesion revascularization | 12 months
  repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion

SECONDARY OUTCOMES:
Angiographic success | 10 minutes after percutaneous transluminal coronary angioplasty
  residual stenosis <50%, TIMI FLOW 3
procedural success | up to 48 hours
  angiographic success in absence of in-hospital events
major adverse cardiac events | 6, 12, 24 and 36 months
  cardiac death, Acute myocardial infarction, target lesion revascularization
very single component of major adverse cardiac events | 6, 12, 24 and 36 months
  cardiac death, Acute myocardial infarction, target lesion revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Bernardo Cortese, Principal Investigator — Clinica San Carlo, Paderno Dugnano, MI, Italy; Antonio Colombo, Study Chair — Humanitas Research Hospital, Rozzano, MI, Italy
Locations (1):
- Unita' Operativa di Cardiologia, Milan, Italy

REFERENCES:
- [Derived] Cortese B, Testa L, Heang TM, Ielasi A, Bossi I, Latini RA, Lee CY, Perez IS, Milazzo D, Caiazzo G, Tomai F, Benincasa S, Nuruddin AA, Stefanini G, Buccheri D, Seresini G, Singh R, Karavolias G, Cacucci M, Sciahbasi A, Ocaranza R, Menown IBA, Torres A, Sengottvelu G, Zanetti A, Pesenti N, Colombo A; EASTBOURNE Investigators. Sirolimus-Coated Balloon in an All-Comer Population of Coronary Artery Disease Patients: The EASTBOURNE Prospective Registry. JACC Cardiovasc Interv. 2023 Jul 24;16(14):1794-1803. doi: 10.1016/j.jcin.2023.05.005. PMID 37495352